CLINICAL TRIAL: NCT02332837
Title: Interactive Tool for Informed Consent: A Randomized Controlled Trial
Brief Title: Interactive Tool for Informed Consent
Acronym: I-TIC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not funded
Sponsor: ThinkWell (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ThinkWell PLOT-03
Record Dates: First submitted 2015-01-04; First posted 2015-01-07 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Informed Consent
Keywords: informed consent, public led trials, shared decision making,

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Digital informed consent (Experimental): Traditional digitally signed text based informed consent
  Intervention A: questionnaire accuracy Intervention B: Questionnaire speed of completion Intervention C: Questionnaire completion rate
  Interventions: Behavioral: Intervention A: Questionnaire accuracy; Behavioral: Intervention B: Questionnaire speed of completion; Behavioral: Intervention C: Questionnaire Completion rate
- Multi-media informed consent (Experimental): Informed consent with images, text and auditory presentation
  Intervention A: questionnaire accuracy Intervention B: Questionnaire speed of completion Intervention C: Questionnaire completion rate
  Interventions: Behavioral: Intervention A: Questionnaire accuracy; Behavioral: Intervention B: Questionnaire speed of completion; Behavioral: Intervention C: Questionnaire Completion rate
- Test to train informed consent (Experimental): Informed consent with images, text, auditory presentation and test to train feature where participants get feedback on comprehension responses throughout the consent and can change them
  Intervention A: questionnaire accuracy Intervention B: Questionnaire speed of completion Intervention C: Questionnaire completion rate
  Interventions: Behavioral: Intervention A: Questionnaire accuracy; Behavioral: Intervention B: Questionnaire speed of completion; Behavioral: Intervention C: Questionnaire Completion rate

INTERVENTIONS:
Behavioral: Intervention A: Questionnaire accuracy — Participants will be tested by questionnaire to measure how well consent is understood
Behavioral: Intervention B: Questionnaire speed of completion — Time to complete questionnaire from time of presentation
Behavioral: Intervention C: Questionnaire Completion rate — Number of participants who complete the questionnaire

SUMMARY:
Online trials require informed consent from participants. Massive online trials make face-to-face signed consent unrealistic and existing consent comprehension could be improved to increase participant safety and understanding.

This trial will compare understanding of traditional digital consent with multi-media consent and with consent that is multi-media and interactive and uses a test and train model.

The computer will assign participants to 1 of 3 methods to present online consent to participants

DETAILED DESCRIPTION:
Online trials require informed consent from participants. Massive online trials make face-to-face signed consent unrealistic and existing consent comprehension could be improved to increase participant safety.

Without accurate knowledge decision-making is not informed. Informed consent for participation in research is part of this process. In online trials the opportunity for face-to-face signed consent with researchers is not an option.

Consent acts as a safeguard that full disclosure occurred. Adequate documentation is evidence against false reports of coercion.

Informed consent inclusive of signed participant information sheets provide a record between researcher and participant of the roles and agreements they share.

According to existing research, only 6% of consents and participant information sheets are written below an eighth grade level of comprehension; 54% of participants with an 8th grade level education partially understood the consent with figures rising to 72% for participants with greater than 8th grade educations, however no participant fully understood the consent materials. The deficits ranged from misunderstandings about risk, side effects, adverse effects reporting, a participants right to withdraw, confidentiality and even the purpose of the trial.

This trial will compare understanding of traditional digital consent with multi-media consent and with consent that is multi-media and interactive and uses a test and train model.

The computer will assign participants to 1 of 3 methods to present online consent to participants

ELIGIBILITY:
Inclusion Criteria:

* pre-screened as eligible for a ThinkWell PLOT trial
* 18 years of age
* No personal email address

Exclusion Criteria:

* not pre-screened or eligible for an existing ThinkWell PLOT trial
* people without internet access
* People who cannot read
* People without the ability to understand the website and informed consent documents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
level of consent comprehension | immediately following intervention
  assessed by accuracy on scored questionnaire

SECONDARY OUTCOMES:
Time to complete consent | immediately following intervention
  Time between presentation of consent materials and signing of consent
Compliance | immediately following intervention
  number of participants who complete consent questionnaire

REFERENCES:
- [Background] Ryan RE, Prictor MJ, McLaughlin KJ, Hill SJ. Audio-visual presentation of information for informed consent for participation in clinical trials. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD003717. doi: 10.1002/14651858.CD003717.pub2. PMID 18254029
- [Background] Gillies K, Huang W, Skea Z, Brehaut J, Cotton S. Patient information leaflets (PILs) for UK randomised controlled trials: a feasibility study exploring whether they contain information to support decision making about trial participation. Trials. 2014 Feb 18;15:62. doi: 10.1186/1745-6215-15-62. PMID 24548781
- [Background] Antoniou EE, Draper H, Reed K, Burls A, Southwood TR, Zeegers MP. An empirical study on the preferred size of the participant information sheet in research. J Med Ethics. 2011 Sep;37(9):557-62. doi: 10.1136/jme.2010.041871. Epub 2011 Apr 8. PMID 21478421
- [Background] Rowbotham MC, Astin J, Greene K, Cummings SR. Interactive informed consent: randomized comparison with paper consents. PLoS One. 2013;8(3):e58603. doi: 10.1371/journal.pone.0058603. Epub 2013 Mar 6. PMID 23484041